CLINICAL TRIAL: NCT00716898
Title: Pharmacokinetics of Low Molecular Weight Heparin in Cancer Patients Compared to Patients With Unstable Angina Pectoris; The Possible Role of Heparanase
Brief Title: Pharmacokinetics of Low Molecular Weight Heparin in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, yair plesser, study manager, Shaare Zedek Medical Center
Other Study IDs: Nasser-2008-1CTIL
Record Dates: First submitted 2008-07-09; First posted 2008-07-16 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Cancer; Thrombosis; Angina Pectoris
Keywords: Condition; Cancer; Patients; Thrombosis; Unstable; Angina; Pectoris
MeSH Terms: conditions — Neoplasms; Thrombosis; Angina Pectoris; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: A. Patients with pathologically or cytologically confirmed diagnosis of advanced solid malignancy.
  B. Venous thromboembolism: Deep vein thrombosis (DVT) confirmed by Doppler ultrasound, or pulmonary embolism confirmed by lung ventilation perfusion scan, or computerized tomography.
  C. Treatment with therapeutic dose of low molecular weight heparin. D. No major surgery during the last month before investigation. E. No evidence of major infectious disease. F. Serum creatinine level < 1.5 mg/dl. G. Informed consent
- 2: A. Patients with unstable angina pectoris/ atypical chest pain, with no evidence of acute myocardial infarction.
  B. Treatment with therapeutic dose of low molecular weight heparin. C. No evidence of VTE. D. No major surgery during the last month before investigation. E. No evidence of major infectious disease. F. No history of malignancy. G. Serum creatinine level < 1.5 mg/dl. H. Informed consent

SUMMARY:
The purpose of the study is to determine the Pharmacokinetics of Low Molecular Weight Heparin (LMWH) in Cancer patients, and compare it to the Pharmacokinetics of LMWH in Patients without cancer. We also intend to detect any correlation between heparanase blood and urine levels and the Pharmacokinetics of LMWH.

DETAILED DESCRIPTION:
Scientific background. The increased risk for venous thromboembolism (VTE) in cancer has long been recognized (1). Since first described by Trousseau in 1865, many aspects of this complex relationship are still obscure (2). Cancer patients have an increased risk for developing thrombosis. Similarly, patients presenting with idiopathic VTE are considered to have a higher risk of developing cancer (3). Approximately 10% of patients with idiopathic VTE harbor an underlying malignancy that can be detected by an extensive diagnostic work-up (4). Clinical data indicate that cancer alone is associated with a 4.1- fold risk of thrombosis, and chemotherapy increases the risk to 6.1- folds (5). Cancer patients develop postoperative VTE at least 2- folds more than patients without cancer undergoing the same surgical procedure (6). Treatment of VTE involves the administration of heparin, low molecular weight heparin (LMWH) or coumarin derivatives. Beside its anticoagulant effects, LMWH may also have an anti-tumoral effect (7-12). The use of LMWH relative to coumarin derivatives was associated with improved survival in patients with solid tumors who did not have metastatic disease at the time of an acute VTE (9). Moreover, addition of LMWH to chemotherapy increased survival of patients with small cell lung cancer (10).

Heparan sulfate proteoglycans (HSPGs) are ubiquitous macromolecules associated with the cell surface and extracellular matrix (ECM) of a wide range of cells of vertebrate and invertebrate tissues. Heparin is structurally related to heparan sulfate (HS), but has higher N- and O-sulfate contents (13). Mammalian endoglycosidase, capable of partially depolymerizing HS chains and commonly referred to as heparanase, has been identified in a variety of cell types and tissues, primarily cancer cells, activated cells of the immune system, platelets, and placenta (14-17). Heparanase is synthesized as a latent 65 kDa precursor whose activation involves proteolytic cleavage at two potential sites located at the N-terminal region of the molecule (Glu109 -Ser110 and Gln157 -lys158), resulting in the formation of two protein subunits that heterodimerize and form the active heparanase enzyme (18). Expression of heparanase correlates with the metastatic potential of human tumor cells (14-16, 19). Furthermore, elevated levels of heparanase were detected in the urine of some patients with aggressive metastatic disease (20). Heparin, LMWH, non-anticoagulant and chemically modified species of heparin (21, 22), as well as other polysaccharides (23, 24) which inhibit experimental metastasis, also inhibit tumor cell heparanase, while other related compounds had a small or no effect on both parameters (21-24). Recently, we demonstrated that the anticoagulant activities of heparin and LMWH can be neutralized by their pre-incubation with heparanase. Transgenic mice overexpressing heparanase, exhibited a hyper-coagulable phenotype expressed by a markedly shorter base-line APTT compared to control mice (25). These results may suggest that resistance to heparin, described in patients with malignancies (26, 27), could be attributed, in part, to high levels of heparanase often observed in cells (28, 29) and body fluids (20) of patients with an aggressive malignant disease. Degradation of heparin and LMWH by heparanase in vivo may be relevant in situations in which heparanase is over-expressed, and treatment with heparin or LMWH is needed (e.g., deep venous thrombosis in patients with pancreatic carcinoma) (29, 30). The pharmacokinetics of LMWH (i.e. the time course of absorption, distribution, metabolism, and degradation) as reflected by its effects upon factor Xa activity, was elucidated in several subgroups of patients (e.g. patients with renal failure, pregnant women…), but to the best of our knowledge was not addressed in patients with advanced solid tumors.

Objectives & expected significance. In view of the above described biological significance of the heparanase enzyme, and taking into account our recent in vitro and in vivo results (heparanase capability to cleave heparin and LMWH; and the altered coagulation profile in transgenic mice overexpressing heparanase) (25), we propose to focus on the following specific aims:

I) Measure plasma and urine heparanase levels in patients with advanced cancer suffering from VTE, and compare it to controls without cancer.

II) Elucidate the pharmacokinetics of LMWH in patients with advanced solid tumors (AST) suffering from VTE, and compare it to the pharmacokinetics of LMWH in patients with unstable angina pectoris.

III) Determine the correlation between heparanase blood levels and the pharmacokinetics of LMWH, if any.

References

1. Rickles FR. Mechanisms of cancer-induced thrombosis in cancer. Pathophysiol Haemost Thromb. 2006; 35: 103-110.
2. Trousseau A: Phlegmasia alba dolens, in: Clinique Medicale de l'Hotel Dieu de Paris. Vol 3, ed 2. Balliere, Paris, 1865; pp 654-712.
3. Valente M, Ponte E. Thrombosis and cancer. Minerva Cardioangiol. 2000; 48: 117-127.
4. Prandoni P. Cancer and venous thromboembolism. Clinical implications of strong association. Pathophysiol Haemost Thromb. 2006; 35: 111-115.
5. Heit JA, Silverstein MD, Mohr DN, Petterson TM, O'Fallon WM, Melton LJ 3rd. Risk factors for deep vein thrombosis and pulmonary embolism: a population-based case-control study. Arch Intern Med. 2000; 160: 809-815.
6. Rickles FR, Levine MN. Epidemiology of thrombosis in cancer. Acta Haematol. 2001; 106: 6-12.
7. von Tempelhoff GF, Harenberg J, Niemann F, Hommel G, Kirkpatrick CJ, Heilmann L. Effect of low molecular weight heparin (Certoparin) versus unfractionated heparin on cancer survival following breast and pelvic cancer surgery: A prospective randomized double-blind trial. Int J Oncol. 2000; 16: 815-824.
8. Kakkar AK, Levine MN, Kadziola Z, Lemoine NR, Low V, Patel HK, Rustin G, Thomas M, Quigley M, Williamson RC. Low molecular weight heparin, therapy with dalteparin, and survival in advanced cancer: the fragmin advanced malignancy outcome study (FAMOUS). J Clin Oncol. 2004; 10: 1944-1948.
9. Lee AY, Rickles FR, Julian JA, Gent M, Baker RI, Bowden C, Kakkar AK, Prins M, Levine MN. Randomized comparison of low molecular weight heparin and coumarin derivatives on the survival of patients with cancer and venous thromboembolism. J Clin Oncol. 2005; 23: 2123-2129.
10. Altinbas M, Coskun HS, Er O, Ozkan M, Eser B, Unal A, Cetin M, Soyuer S. A randomized clinical trial of combination chemotherapy with and without low-molecular-weight heparin in small cell lung cancer. J Thromb Haemost. 2004; 2: 1266-1271.
11. Klerk CP, Smorenburg SM, Otten HM, Lensing AW, Prins MH, Piovella F, Prandoni P, Bos MM, Richel DJ, van Tienhoven G, Buller HR. The effect of low molecular weight heparin on survival in patients with advanced malignancy. J Clin Oncol. 2005; 23: 2130-2135.
12. Meyer G, Marjanovic Z, Valcke J, Lorcerie B, Gruel Y, Solal-Celigny P, Le Maignan C, Extra JM, Cottu P, Farge D. Comparison of low-molecular-weight heparin and warfarin for the secondary prevention of venous thromboembolism in patients with cancer: a randomized controlled study. Arch Intern Med. 2002; 162:1729-1735.
13. Casu B, Lindahl U. Structure and biological interactions of heparin and heparan sulfate. Adv Carbohydr Chem Biochem. 2001; 57: 159-206.
14. Parish CR, Freeman C, Hulett MD. Heparanase: a key enzyme involved in cell invasion. Biochim Biophys Acta. 2001; 1471: M99-108.
15. Vlodavsky I, Friedmann Y. Molecular properties and involvement of heparanase in cancer metastasis and angiogenesis. J Clin Invest. 2001; 108: 341-347.
16. Nakajima M, Irimura T, Nicolson GL. Heparanases and tumor metastasis. J Cell Biochem. 1988; 36:157-167.
17. Dempsey LA, Brunn GJ, Platt JL. Heparanase, a potential regulator of cell-matrix interactions. Trends Biochem Sci. 2000; 25: 349-351.
18. Levy-Adam F, Miao HQ, Heinrikson RL, Vlodavsky I, Ilan N. Heterodimer formation is essential for heparanase enzymatic activity. Biochem Biophy Res Commun. 2003; 308: 885-891.
19. Vlodavsky I, Friedmann Y, Elkin M, Aingorn H, Atzmon R, Ishai-Michaeli R, Bitan M, Pappo O, Peretz T, Michal I, Spector L, Pecker I. Mammalian heparanase: gene cloning, expression and function in tumor progression and metastasis. Nat Med. 1999; 5: 793-802.
20. Shafat I, Zchria E, Nisman B, Nadir Y, Nakhoul F, Vlodavsky I, Ilan N. An ELISA method for the detection and quantification of human heparanase. Biochem Biophy Res Commun. 2006; 341: 958-963.
21. Vlodavsky I, Mohsen M, Lider O, Svahn CM, Ekre HP, Vigoda M, Ishai-Michaeli R, Peretz T. Inhibition of tumor metastasis by heparanase inhibiting species of heparin. Invasion Metastasis. 1994; 14: 290-302.
22. Parish CR, Coombe DR, Jakobsen KB, Bennett FA, Underwood PA. Evidence that sulphated polysaccharides inhibit tumour metastasis by blocking tumour-cell-derived heparanases. Int J Cancer. 1987; 40: 511-518.
23. Parish CR, Freeman C, Brown KJ, Francis DJ, Cowden WB. Identification of sulfated oligosaccharide-based inhibitors of tumor growth and metastasis using novel in vitro assays for angiogenesis and heparanase activity. Cancer Res. 1999; 59: 3433-3441.
24. Miao HQ, Elkin M, Aingorn E, Ishai-Michaeli R, Stein CA, Vlodavsky I. Inhibition of heparanase activity and tumor metastasis by laminarin sulfate and synthetic phosphorothioate oligodeoxynucleotides. Int J Cancer. 1999; 83: 424-431.
25. Nasser NJ, Sarig G, Brenner B, Nevo E, Goldshmidt O, Zcharia E, Li JP, Vlodavsky I. Heparanase neutralizes the anticoagulation properties of heparin and low-molecular-weight heparin. J Thromb Haemost. 2006; 4: 560-565.
26. Levy JH. Heparin resistance and antithrombin: should it still be called heparin resistance? Journal of cardiovascular anesthesia. 2004; 18: 129-130.
27. Deitcher SR. Cancer and thrombosis: mechanisms and treatment. J Thromb Thrombolysis. 2003; 16: 21-31.
28. Gohji K, Hirano H, Okamoto M, Kitazawa S, Toyoshima M, Dong J, Katsuoka Y, Nakajima M. Expression of three extracellular matrix degradative enzymes in bladder cancer. Int J Cancer. 2001; 95: 295-301.
29. Koliopanos A, Friess H, Kleeff J, Shi X, Liao Q, Pecker I, Vlodavsky I, Zimmermann A, Buchler MW. Heparanase expression in primary and metastatic pancreatic cancer. Cancer Res. 2001; 61: 4655-59.
30. Kim AW, Xu X, Hollinger EF, Gattuso P, Godellas CV, Prinz RA. Human heparanase-1 gene expression in pancreatic adenocarcinoma. J Gastrointest Surg. 2002; 6: 167-172.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with therapeutic dose of low molecular weight heparin
* Serum creatinine level < 1.5 mg/dl.

Exclusion Criteria:

* major surgery during the last month before investigation
* evidence of major infectious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated at SZMC
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2009-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Low Molecular Weight Heparin (LMWH) in Cancer patients | Interim analysis and at the end of the trial

SECONDARY OUTCOMES:
The role of heparanase on the Pharmacokinetics of Low Molecular Weight Heparin (LMWH) in Cancer patients | End of the study

CONTACTS AND LOCATIONS:
Overall Officials: Nicola j nasser, MD, PhD, Principal Investigator — Shaare Zedek MC
Locations (1):
- Shaare Zedek Medicla Center, Jerusalm, Israel, Israel

REFERENCES:
- [Derived] Nasser NJ, Na'amad M, Weinberg I, Gabizon AA. Pharmacokinetics of low molecular weight heparin in patients with malignant tumors. Anticancer Drugs. 2015 Jan;26(1):106-11. doi: 10.1097/CAD.0000000000000176. PMID 25280062